CLINICAL TRIAL: NCT03570164
Title: Comparison of Vasodilative Effects Between Sevoflurane and Desflurane Using Peripheral Perfusion Index
Brief Title: Hemodynamics for Equi-MAC Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kangbuk Samsung Hospital (Other)
Responsible Party: Principal Investigator, Kyoung-Ho Ryu, MD, Assistant professor, Kangbuk Samsung Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2018-05-019
Record Dates: First submitted 2018-06-15; First posted 2018-06-26 (Actual); Last update posted 2019-10-21 (Actual); Status verified 2019-10

CONDITIONS: Anesthesia
MeSH Terms: interventions — Sevoflurane; Desflurane

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sevoflurane (Experimental): Anesthesia is maintained with sevoflurane.
  Interventions: Drug: Sevoflurane
- Desflurane (Experimental): Anesthesia is maintained with desflurane.
  Interventions: Drug: Desflurane

INTERVENTIONS:
Drug: Sevoflurane — End-tidal concentration of sevoflurane is maintained at age-corrected 1.0 minimum alveolar concentration throughout the study period.
  Other Names: Sevorane
  Arms: Sevoflurane
Drug: Desflurane — End-tidal concentration of desflurane is maintained at age-corrected 1.0 minimum alveolar concentration throughout the study period.
  Other Names: Suprane
  Arms: Desflurane

SUMMARY:
The aim of this study is to compare the peripheral perfusion index values produced by equi-MAC of sevoflurane and desflurane in patients undergoing single-agent inhalation anesthesia.

DETAILED DESCRIPTION:
Ether derivative anesthetics, including sevoflurane and desflurane, have direct activity on vascular tissue and both are vasodilators. However, there has been no direct comparison of vasodilative effect between sevoflurane and desflurane in vivo in humans. Peripheral perfusion index derived from photoplethysmographic waveform reflects peripheral vasomotor tone. Therefore, the purpose of this study is to compare the peripheral perfusion index values produced by sevoflurane and desflurane at equipotent concentration in patients undergoing single-agent inhalation anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* patients aged between 19 and 65 yr
* patients with American Society of Anesthesiologists physical status classification I or II
* patients scheduled for elective arthroscopic knee surgery under general anesthesia
* patients obtaining written informed consent

Exclusion Criteria:

* patients with a history of any disease associated with the autonomic nervous system
* patients receiving any medication affecting the sympathetic or parasympathetic nervous systems
* patients with cardiac arrhythmia, diabetes mellitus, and alcohol or drug abuse
* pregnant women

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2018-06-18 (Actual); Primary Completion 2018-11-13 (Actual); Study Completion 2018-11-13 (Actual)

PRIMARY OUTCOMES:
peripheral perfusion index | After a 30-min waiting period from the induction of anesthesia
  peripheral perfusion index value at a steady-state anesthesia of age-corrected 1.0 MAC

SECONDARY OUTCOMES:
mean arterial pressure | After a 30-min waiting period from the induction of anesthesia
  mean arterial pressure at a steady-state anesthesia of age-corrected 1.0 MAC
heart rate | After a 30-min waiting period from the induction of anesthesia
  heart rate at a steady-state anesthesia of age-corrected 1.0 MAC

CONTACTS AND LOCATIONS:
Overall Officials: Kyoung-Ho Ryu, M.D., Principal Investigator — Kangbuk Samsung Hospital
Locations (1):
- Kangbuk Samsung Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ryu KH, Hwang SH, Shim JG, Ahn JH, Cho EA, Lee SH, Byun JH. Comparison of vasodilatory properties between desflurane and sevoflurane using perfusion index: a randomised controlled trial. Br J Anaesth. 2020 Dec;125(6):935-942. doi: 10.1016/j.bja.2020.07.050. Epub 2020 Sep 18. PMID 32958203